CLINICAL TRIAL: NCT04723667
Title: Effects of an Empowerment-based Psycho-behavioral Program on Neuropsychiatric Symptoms, Cognitive Function and Health-related Quality of Life of Persons With Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: Effects of an Empowerment-based Psycho-behavioral Program on Persons With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Rose Sin Yi Lin, PhD student, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2020-12-14; First posted 2021-01-26 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment
Keywords: neuropsychiatric symptoms; randomized controlled trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This study aims to evaluate the effects of a 13-week empowerment-based psycho-behavioral program to improve neuropsychiatric symptoms, cognitive functions, and health-related quality of life among persons with mild cognitive impairment. A feasibility pilot study will be first evaluated in a pilot study among 30 participants with MCI and subsequently a full-scale randomized controlled trial will be conducted.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors were blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 13-week multimodal intervention
  Interventions: Behavioral: 13-week multimodal intervention
- Active control (Active Comparator): 5-week health education programme
  Interventions: Behavioral: 5-week health education programme

INTERVENTIONS:
Behavioral: 13-week multimodal intervention — The experimental intervention was a 13-week multimodal intervention consists of five-weekly, 90-minute, face-to-face sessions to be delivered in a group format (six to eight participants per group), followed by two weekly and three biweekly telephone follow-ups. The five face-to-face sessions covered brain health information, booster memory power, reducing stressors, optimizing strength and active lifestyle engagement.
  Arms: Intervention
Behavioral: 5-week health education programme — The health education program consisted of three topics (fall prevention, oral care and home hygiene), with two tele-booster follow up
  Arms: Active control

SUMMARY:
This study aims to evaluate the effects of a 13-week empowerment-based psycho-behavioral program to improve neuropsychiatric symptoms, cognitive functions, and health-related quality of life among persons with mild cognitive impairment. Its feasibility will be first evaluated in a pilot study and subsequently in a randomized controlled trial (RCT)

DETAILED DESCRIPTION:
Dementia has become a global pandemic. It affects 50 million people worldwide and this number is projected to have a three-fold increase to over 150 million by 2050. Dementia is characterized by a progressive deterioration in cognitive functions that interferes an individual to live independently. It jeopardizes the quality of life of the sufferers and their families and poses tremendous economic burden on health and social systems. In 2018, the total cost incurred by dementia worldwide was up to US$ 1 billion and it was forecasted to double in 2050. Since dementia is incurable, efforts to mitigate the burgeoning population of dementia should be directed to its prodromal reversible stage, that is, mild cognitive impairment (MCI).

MCI refers to the transitional stage between normal age-related cognitive decline and dementia. It is characterized by cognitive decline in a single or multiple cognitive domains including memory, executive functions, attention, language and visuospatial skills, but the ability to engage in activities of daily living is preserved. The global prevalence of MCI is 10 to 20% in persons aged 65 or older, and up to 25.9% for those aged above 80 years.

Current research effort focuses on addressing the cognitive symptoms of persons with MCI (PwMCI), least attention was paid to the co-existing neuropsychiatric symptoms (NPS). Such non-cognitive symptoms, indeed, affect persons in different stages of cognitive impairment, there is no exception for MCI. NPS is an umbrella term that captures psychological and behavioural symptoms, typical psychological symptoms encompass depression, apathy, and anxiety, which may cluster into a syndrome and precipitate behavioural symptoms such as agitation and disinhibition. Two systematic reviews simultaneously reported that up to 85% of the MCI population are afflicted with at least one of these symptoms, with depression being the most prevalent followed by anxiety and irritability. Comparing to those without such symptoms, they tend to have poorer quality of life, more severe functional loss, and with a fourfold increased risk for progression to dementia.

Despite the fact NPS is highly prevalence among PwMCI, effective management with comprehensive outcome measurement is yet to be determined. An empowerment-based, comprehensive multimodal intervention with MCI-specific outcome measurement on overall NPS is warranted. Such intervention should cover skills compensation with transferral into daily life, lifestyle reform, strength-based activity, cognitive restructuring, and disease-specific education. This study aims to evaluate an empowerment-based psycho-behavioral program on improving NPS, cognitive function and health-related quality of life among persons with MCI. This is a mix-methods study comprising an assessor-blinded randomized controlled trial and a descriptive qualitative study

As for the sample size calculation, the sample size of the pilot study was set based on a general rule of thumb of 30 participants, which has been shown adequate for exploring feasibility and outcome estimates to inform future trials. Those for the major study, Power analysis using G*Power was performed to estimate the sample size for the RCT. According to the result of a systematic review that the pooled effect size of the non-pharmacological interventions on depression among persons with MCI was 0.47 (Lin et al., 2020), this study conservatively assumed the effect size of a similar but more comprehensive intervention on the primary outcome of NPS as 0.4. A sample size of 125 per study group is needed to achieve 80% power at a 5% level of significance, allowing a 20% attrition for a 17-week study.

Block randomization was used to allocate the participants to an intervention group, which received an empowerment-based psycho-behavioral program, or a control group, which received a health education program, at 1:1 ratio. The random sequence was generated by a computer randomization software on randomization.com. Each number was printed on a standard 2cm x 2cm memo and placed into an opaque and sealed envelope. To assure adequate allocation concealment, the allocation procedure was conducted by an independent research assistant who was not involved in this study.

For the quantitative data, all test comparisons were set at two-side at a level of significance of 0.05. The quantitative data were analyzed by SPSS Statistics (version 27) according to the intention-to-treat principle. Descriptive statistics were used to summarize the socio-demographic data, clinical profile, and outcome variables. The similarity of study groups at baseline was examined using chi-square test for categorical data and independent t-test for continuous data. All participants were assessed at baseline (T0), immediate post-test (T1), and four-week post-test (T2) to determine changes in their MBI-C, GDS-SF, AES, K10, HK-MoCA, MIC, and SF-12v2 scores. A generalized estimating equation (GEE) model was used to determine between- and within-group differences in outcome variables across three data collection timepoints. All statistical analyses were two-tailed with a 5% level of statistical significance. Effect size estimates were calculated for all mean differences using Cohen's d values, and were classified as negligible (d<0.2), small (0.2≤ d<0.5), medium (0.5≤d< 0.8), or large (d≥0.8) effects (Lakens, 2013). Post-hoc power analysis was performed for all outcome variables using G*Power software. Individual semi-structured interviews were conducted to explore the perceived effects of the psycho-behavioral program and the qualitative data were analyzed by content analysis.

Lin, R. S. Y., Yu, D. S. F., Chau, P. H., & Li, P. W. C. (2021). An empowerment-psycho-behavioral program on neuropsychiatric symptoms in persons with mild cognitive impairment: Study protocol of a randomized controlled trial. Journal of Advanced Nursing.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 years old or above
2. Able to communicate in Cantonese
3. Diagnosis with MCI as defined by the following criteria:

I. Presence of significant cognitive complaints as reflected by self-report II. Abnormal objective cognitive performance defined as < 1.5 standard deviations from age and education matched normal persons on Hong Kong Chinese version of Montreal Cognitive Assessment (HK-MoCA), which is a 12-item instrument measuring cognitive functions, more details are outlined under the session of outcome measures III. Independence in daily living as evaluated through clinical interviews

Exclusion Criteria:

1. With the confirmed diagnosis of any forms of dementia
2. With the confirmed diagnosis of psychiatric morbidities, or history with stroke, brain injury and other neurological conditions that may affect cognitive, behavioral, and emotional functioning which may confound outcome measurement and limit their participation in the study
3. With hearing or visual impairment that may hinder participation in research activities
4. Current use of any cognitive intervention or electromagnetic stimulation that confound cognitive outcomes

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Mild Behavioral Impairment - Checklist (MBI-C) | 17 weeks
  Mild Behavioral Impairment - Checklist (MBI-C), this 34-item questionnaire will be used to measure five domains of NPS, including decreased motivation, emotional dysregulation, impulse dyscontrol, social inappropriateness, and abnormal perception or thought content.
Kessler Psychological Distress Scale (K10) | 17 weeks
  Kessler Psychological Distress Scale (K10), this 10-item instrument will be used to measure the level of non-specific psychological distress, primarily anxiety and depression, over the past month on a '1-5' 5-point Likert scale.
Apathy Evaluation Scale (AES-S) | 17 weeks
  Apathy Evaluation Scale (AES-S), this 18-item instrument will be used to measure apathy over the past four weeks on a '1-4' 4-point Likert scale.
Geriatric Depression Scale - Short Form (GDS-SF) | 17 weeks
  Geriatric Depression Scale - Short Form (GDS-SF), this 15-item instrument will be used to measure depression.

SECONDARY OUTCOMES:
Hong Kong version of the Montreal Cognitive Assessment (HK-MoCA) | 17 weeks
  Hong Kong version of the Montreal Cognitive Assessment (HK-MoCA), this 12-item instrument will be used to measure cognitive functions including visuospatial functions, naming, verbal memory, abstraction, delay memory, calculation, and orientation.
Memory Inventory in Chinese (MIC) | 17 weeks
  Memory Inventory in Chinese (MIC), this 27-item instrument will be used to measure subjective memory deficit on a 5-point Likert Scale.
Hong Kong Short Form -12 (HK-SF12) | 17 weeks
  Hong Kong Short Form -12 (HK-SF12), this 12-item instrument will be used to measure perceived health-related quality of life including physical and social functioning, physical and emotional role, mental health, bodily pain, general health perception, and vitality

CONTACTS AND LOCATIONS:
Overall Officials: Rose Lin, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Rose Lin, Hong Kong
  - University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Anonymity will be reassured by subject codes without identifiers of the participants. All the data collected will be stored in secure place and can only be accessed by research team members. All the data will be kept for five years and will be destroyed upon the completion of the study as to protect participants' confidentiality.

REFERENCES:
- [Derived] Lin RSY, Yu DSF, Pui Hing Chau P, Li PWC. An empowerment-psycho-behavioral program on neuropsychiatric symptoms in persons with mild cognitive impairment: Study protocol of a randomized controlled trial. J Adv Nurs. 2021 Aug;77(8):3507-3517. doi: 10.1111/jan.14871. Epub 2021 Apr 28. PMID 33909293